CLINICAL TRIAL: NCT02212977
Title: Comparison of Topical Skin Adhesive to Subcuticular Suture Closure of Implantable Port Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00056064
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Port-A-Cath Placement; Octylcyanoacrylate
Keywords: Port Catheter; Octyl 2-cyanoacrylate; 2-octylcyanoacrylate
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suture (Active Comparator): Skin incision closure with standard subcuticular technique using a running 4-0 Polysorb suture
  Interventions: Procedure: Suture
- Octylcyanoacrylate (Experimental): Skin incision closure with topic skin adhesive Octylcyanoacrylate
  Interventions: Device: Octylcyanoacrylate

INTERVENTIONS:
Device: Octylcyanoacrylate — Skin incision closure with topic skin adhesive Octylcyanoacrylate
  Other Names: Octyl 2-cyanoacrylate; 2-octylcyanoacrylate
  Arms: Octylcyanoacrylate
Procedure: Suture — Skin incision closure with standard subcuticular technique using a running 4-0 Polysorb suture
  Arms: Suture

SUMMARY:
Hypothesis is that incision closure with octylcyanoacrylate is inferior to closure with stitches in Port a Cath patients, who, as a population, are at increased risk for complications. All adult patients who present for initial Port a Cath placement during the recruitment period will be eligible to participate in the study. Subjects will be randomized to either skin incision closure with standard stitches or closure with skin glue. Time to complete skin closure and costs of closure will be compared. Patients will be evaluated approximately one month and three months from the procedure to assess for complications of wound breakdown or infection, as well as for the appearance of the Port a Cath incision.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥18 years) who present for initial implantable port placement during the recruitment period will be eligible to participate in the study

Exclusion Criteria:

* Patients who cannot provide informed consent for the procedure will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kim, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suture | Octylcyanoacrylate
Started | 55 | 54
Completed | 50 | 48
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suture | Octylcyanoacrylate | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (7.5) | 58.3 (7.6) | 58.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 35 | 81
  Male | 9 | 19 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complication of Wound Dehiscence
Description: To compare complication rates, including wound dehiscence and infection rates between implantable port incisions closed with topical skin adhesive versus absorbable subcuticular sutures.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Suture | Octylcyanoacrylate
Number analyzed (Participants) | 50 | 48
participants | 0 | 0

2. Primary Outcome: Number of Participants With Complication of Infection
Description: as for outcome 1
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Suture | Octylcyanoacrylate
Number analyzed (Participants) | 50 | 48
participants | 2 | 1

3. Secondary Outcome: Healing-incision Cosmesis Score by Visual Analogue Scale
Description: To compare resultant cosmesis with topic skin adhesive closure versus suture closure. Scale is 1-10 with 1 as the best possible outcome and 10 is the worst possible outcome.
Time Frame: 3 months
Population: Only participants who completed the Healing-incision cosmesis score by Visual Analogue Scale were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suture | Octylcyanoacrylate
Number analyzed (Participants) | 45 | 41
units on a scale | 4.46 (2.4) | 4.4 (2.6)

4. Secondary Outcome: Closure Time
Description: To compare closure time and associated costs between these two methods of skin closure.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suture | Octylcyanoacrylate
Number analyzed (Participants) | 55 | 54
minutes | 8.6 (3.7) | 1.6 (0.8)

5. Secondary Outcome: Closure Materials Cost
Description: Per unit cost for suture and octylcyanoacrylate
Time Frame: Baseline
Measure: Number; unit: dollars
Arm/Group | Suture | Octylcyanoacrylate
Number analyzed (Participants) | 55 | 54
dollars | 2.54 | 25.92

ADVERSE EVENTS:
Arm/Group | Suture | Octylcyanoacrylate
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

LIMITATIONS AND CAVEATS:
Small sample size, underpowered to demonstrate small differences in rates of dehiscence or infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes